CLINICAL TRIAL: NCT03713073
Title: Clinical and Histological Outcomes of Allogenic Amnion Chorion Membrane in the Healing of Free Gingival Graft Donor Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Chun-Teh Lee, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-DB-18-0303
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Palatal Wound

STUDY DESIGN:
Intervention Model Description: The study is a "split-mouth design," in which two treatments (test and control) are randomly assigned to either the right or left halves of the dentition/palate.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Allogenic amnion chorion membrane (Experimental): Allogenic amnion chorion membrane (ACM) is a minimally manipulated allograft amnion chorion tissue for use as a wound covering in dental surgery.
  Interventions: Device: Allogenic amnion chorion membrane
- Collagen dressing (Active Comparator): Collagen dressing is used to cover wounds in dental surgery.
  Interventions: Device: Collagen dressing

INTERVENTIONS:
Device: Allogenic amnion chorion membrane — Allogenic amnion chorion membrane (ACM) is a minimally manipulated allograft amnion chorion tissue for use as a wound covering in dental surgery.
  Arms: Allogenic amnion chorion membrane
Device: Collagen dressing — Collagen dressing is used to cover wounds in dental surgery.
  Arms: Collagen dressing

SUMMARY:
The purpose of this study is to compare an allogenic amnion chorion membrane to a collagen dressing in palatal wound healing after harvesting free gingival graft (FGG).

ELIGIBILITY:
Inclusion Criteria:

* patients attending the Clinic for Graduate Periodontics at The University of Texas health Science Center at Houston School of Dentistry who are in need of a Free Gingival Graft procedure to augment keratinized gingiva, augment ridge, or cover recession defects.
* systemically healthy or with controlled common systemic conditions, such as hypertension, that will not affect wound healing.

Exclusion Criteria:

* size of the FGG that the patient needs bigger than the size of FGGs that have to be harvested in this study (two 8mm (width) x 10mm (length) x ≈1.5mm (thickness) FGG).
* current heavy smokers(>10 cigarettes/day) (patients who stop smoking more than one year are eligible)
* have diabetes or other systemic diseases that may comprise healing
* take antibiotics and/or analgesics within one week before the procedure and have loss of sensation on the palate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Teh Lee, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Lee CT, Umoh EN, Husain A, Gomnam N, Tribble G, Wang BY, Min S. Clinical and histological outcomes of allogenic amnion-chorion membrane for palatal donor site healing. J Periodontol. 2025 Jul 8. doi: 10.1002/jper.11370. Online ahead of print. PMID 40627760

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: palatal wound site
Groups:
- All Participants: The study is a "split-mouth design." For each participant, there were 2 palatal wound sites (one on the right side and one on the left side), and for each participant, allogenic amnion chorion membrane (ACM) was placed on one of the wound sites and collagen dressing was placed on the other wound site. In other words, each participant received both interventions, and the interventions were received at the same time. The side of placement of the two interventions was randomized.
  Allogenic amnion chorion membrane (ACM) is a minimally manipulated allograft amnion chorion tissue for use as a wound covering in dental surgery.
  Collagen dressing is used to cover wounds in dental surgery.
Period: Overall Study
Arm/Group | All Participants
Started | 19; 38 palatal wound site
Allogenic Amnion Chorion Membrane | 19; 19 palatal wound site
Collagen Dressing | 19; 19 palatal wound site
Completed | 19; 38 palatal wound site
Not Completed | 0; 0 palatal wound site

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.55 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Body mass index (BMI) [Count of Participants; unit: Participants]
  18.5-24.9 kg/m² | 13
  25-29.9 kg/m² | 2
  greater than 30 kg/m² | 4
Number of participants with hypertension [Count of Participants; unit: Participants] | 4
Number of participants who currently smoke [Count of Participants; unit: Participants] | 1
Physical status as indicated by American Society of Anesthesiologists (ASA) Class [Count of Participants; unit: Participants] — ASA class I is a normal healthy patient who is non-smoking with no or minimal alcohol use. ASA class II is a patient with mild systemic disease without substantive functional limitations, for instance may be a current smoker, social alcohol drinker, pregnant, or obese (30<BMI<40), or well-controlled diabetes mellitus and hypertension (DM/HTN) or mild lung disease.
  Participants
    ASA class I | 10
    ASA class II | 9

OUTCOME MEASURES:

1. Primary Outcome: Size of Wound Area
Description: The wound area will be assessed by means of a clinical picture. The picture will be taken with an angulation perpendicular to the wound. A periodontal probe will be placed by the wound as a reference scale. Wound area is defined as the area without epithelization. The wound area on the picture will be measured by ImageJ.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
micrometers (μm) | 80 (0) | 80 (0)

2. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
micrometers (μm) | 35.9 (12.2) | 37.3 (12.9)

3. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 10 days
Population: Data for this outcome were not collected for four in the allogenic amnion chorion membrane arm and four in the collagen dressing arm.
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 15 | 15
micrometers (μm) | 22.9 (10.7) | 25.6 (10.2)

4. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 14 days
Population: Data for this outcome were not collected for one in the allogenic amnion chorion membrane arm and one in the collagen dressing arm.
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
micrometers (μm) | 13.3 (9.1) | 14.1 (7.9)

5. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 21 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
micrometers (μm) | 2.8 (3.4) | 4.1 (4.1)

6. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 28 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
micrometers (μm) | 0 (0) | 0.25 (1.0)

7. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 45 days
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
micrometers (μm) | 0 (0) | 0 (0)

8. Primary Outcome: Size of Wound Area
Description: as for outcome 1
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
micrometers (μm) | 0 (0) | 0 (0)

9. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: Epithelialization is measured by means of bubble formation after dripping hydrogen peroxide (3%) to the wound surface. Less bubbles indicate greater epithelialization, and epithelialization will be ranked as total, partial or none.
Time Frame: baseline
Population: Data were not collected at this time point for this outcome measure.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 4 days
Population: Data for this outcome were not collected for one in the allogenic amnion chorion membrane arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 19
Participants
  no epithelialization | 18 | 19
  partial epithelialization | 0 | 0
  total epithelialization | 0 | 0

11. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 10 days
Population: Data for this outcome were not collected for three in the allogenic amnion chorion membrane arm and four in the collagen dressing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 16 | 15
Participants
  no epithelialization | 0 | 0
  partial epithelialization | 15 | 15
  total epithelialization | 1 | 0

12. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 14 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  no epithelialization | 0 | 0
  partial epithelialization | 7 | 7
  total epithelialization | 11 | 11

13. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 21 days
Population: Data for this outcome were not collected for one in the allogenic amnion chorion membrane arm and seven in the collagen dressing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 11
Participants
  no epithelialization | 0 | 0
  partial epithelialization | 1 | 0
  total epithelialization | 17 | 11

14. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 28 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  no epithelialization | 0 | 0
  partial epithelialization | 0 | 0
  total epithelialization | 18 | 18

15. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  no epithelialization | 0 | 0
  partial epithelialization | 0 | 0
  total epithelialization | 19 | 19

16. Secondary Outcome: Number of Participants Stratified as Per the Degree of Epithelialization of Wound
Description: as for outcome 9
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  no epithelialization | 0 | 0
  partial epithelialization | 0 | 0
  total epithelialization | 19 | 19

17. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: The color of wound site will be compared to the adjacent gingiva by using a 4-point scale: 1. Obvious difference; 2. Noticeable difference; 3. Disguisable difference; or 4. No noticeable difference in comparison with adjacent gingiva.
Time Frame: baseline
Population: Data were not collected at this time point for this outcome measure.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  obvious difference | 19 | 19
  noticeable difference | 0 | 0
  disguisable difference | 0 | 0
  no noticeable difference | 0 | 0

19. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 10 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 15 | 15
Participants
  obvious difference | 15 | 15
  noticeable difference | 0 | 0
  disguisable difference | 0 | 0
  no noticeable difference | 0 | 0

20. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 14 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  obvious difference | 5 | 10
  noticeable difference | 12 | 6
  disguisable difference | 1 | 2
  no noticeable difference | 0 | 0

21. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 21 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  obvious difference | 0 | 0
  noticeable difference | 6 | 7
  disguisable difference | 7 | 10
  no noticeable difference | 5 | 1

22. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 28 days
Population: Data for this outcome were not collected for three in the allogenic amnion chorion membrane arm and three in the collagen dressing arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 16 | 16
Participants
  obvious difference | 0 | 0
  noticeable difference | 0 | 2
  disguisable difference | 9 | 12
  no noticeable difference | 7 | 2

23. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 45 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  obvious difference | 0 | 0
  noticeable difference | 0 | 0
  disguisable difference | 4 | 6
  no noticeable difference | 14 | 12

24. Secondary Outcome: Relative Difference in Color of Wound Site Compared to Adjacent Gingiva
Description: as for outcome 17
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  obvious difference | 0 | 0
  noticeable difference | 0 | 0
  disguisable difference | 2 | 3
  no noticeable difference | 17 | 16

25. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: baseline
Population: Data were not collected at this time point for this outcome measure.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 19 | 19

27. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 18 | 19

28. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 18 | 18

29. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 19 | 19

30. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 19 | 19

31. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 19 | 19

32. Secondary Outcome: Number of Participants With Haemostasis of Wound Area
Description: Haemostasis is achieved when no bleeding of the wound site is actively seen.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants | 19 | 19

33. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: Pain will be assessed by a Visual Analogue Scale (VAS). Scores range form 0 to 10. 0 indicates no pain, 1 indicates minimal pain, and 10 indicates severe pain.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 7.89 (2.13) | 7.89 (2.13)

34. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 4.42 (1.57) | 4.42 (1.57)

35. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 1.63 (2.31) | 1.63 (2.31)

36. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 0.53 (1.26) | 0.53 (1.26)

37. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 0.32 (1.00) | 0.32 (1.00)

38. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 0 (0) | 0 (0)

39. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 45 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 0 (0) | 0 (0)

40. Secondary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 33
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
units on a scale | 0 (0) | 0 (0)

41. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: Sensibility will be assessed with a periodontal probe using a rubbing movement and pin-pressure nociception. Patients will be asked to rate their sensitivity based on a 3-point verbal descriptor scale (VDS): no loss of sensation, mild/moderate loss of sensation, or severe loss of sensation.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  no loss of sensation | 19 | 19
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

42. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: Sensibility will be assessed with a periodontal probe using a rubbing movement and pin-pressure nociception. Patients will be asked to rate their sensibility based on a 3-point verbal descriptor scale (VDS): no loss of sensation, mild/moderate loss of sensation, or severe loss of sensation.
Time Frame: 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  no loss of sensation | 19 | 19
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

43. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: as for outcome 42
Time Frame: 10 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 15 | 15
Participants
  no loss of sensation | 15 | 15
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

44. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: as for outcome 42
Time Frame: 14 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  no loss of sensation | 18 | 18
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

45. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: as for outcome 42
Time Frame: 21 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  no loss of sensation | 18 | 18
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

46. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: as for outcome 42
Time Frame: 28 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
Participants
  no loss of sensation | 18 | 18
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

47. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: as for outcome 42
Time Frame: 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  no loss of sensation | 19 | 19
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

48. Secondary Outcome: Sensibility of the Wound Area as Indicated by Number of Participants Who Lost Sensation as Assessed by a 3-point Verbal Descriptor Scale (VDS)
Description: as for outcome 42
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
Participants
  no loss of sensation | 19 | 19
  mild/moderate loss of sensation | 0 | 0
  severe loss of sensation | 0 | 0

49. Secondary Outcome: Volume of Wound
Description: The wound area will analyzed with an intraoral scanner, and three-dimensional images will be reconstructed to determine the volume of the wound.
Time Frame: baseline
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 4 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 10 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 14 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 21 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 28 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 45 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Volume of Wound
Description: as for outcome 49
Time Frame: 60 days
Population: There is not enough usable data collected for any participant to summarize and report this outcome measure accurately.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Clinician's Feedback on the Wound Dressing Material as Assessed by a Questionnaire
Time Frame: at the time of placement of the wound dressing material
Population: Data for this outcome measure were not collected.
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Number of Neutrophil Cells as Assessed by Light Microscopy of Haematoxylin and Eosin (H&E)-Stained Biopsy Sections
Description: Gingival specimen biopsies (4mm in diameter, 1.5mm in thickness) will be harvested. The histological sections will be evaluated using a Nikon light microscope.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: neutrophil cells
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
neutrophil cells | 62.1 (29.9) | 65 (22.6)

59. Secondary Outcome: Number of Neutrophil Cells as Assessed by Light Microscopy of Haematoxylin and Eosin (H&E)-Stained Biopsy Sections
Description: as for outcome 58
Time Frame: 10 days
Population: Data for this outcome were not collected for one in the allogenic amnion chorion membrane arm and two in the collagen dressing arm.
Measure: Mean (Standard Deviation); unit: neutrophil cells/field
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 17
neutrophil cells/field | 80 (47.7) | 88 (35.8)

60. Secondary Outcome: Change in Percentage of Collagen Density in Wound Area as Assessed by Light Microscopy of Masson's Trichrome-stained Biopsy Sections
Time Frame: baseline, 10 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of collagen density
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 18
percentage of collagen density | 1.15 (2.41) | 3.38 (2.63)

61. Secondary Outcome: Thickness of the Epithelium as Assessed by Light Microscopy of Haematoxylin and Eosin (H&E)-Stained Biopsy Sections
Description: Gingival specimen biopsies (4mm in diameter, 1.5mm in thickness) will be harvested. The histological sections will be evaluated using a Nikon light microscope, and Nikon NIS-Elements Advanced Research (AR) Imagine Software will be used to calculate the thickness of the epithelium.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
micrometers (μm) | 302.2 (95.2) | 291 (79.7)

62. Secondary Outcome: Thickness of the Epithelium as Assessed by Light Microscopy of Haematoxylin and Eosin (H&E)-Stained Biopsy Sections
Description: as for outcome 61
Time Frame: 10 days
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: micrometers (μm)
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 17
micrometers (μm) | 339.6 (94.4) | 339.3 (118.6)

63. Secondary Outcome: Angiogenesis as Indicated by Number of Blood Vessels as Assessed by Light Microscopy of Biopsy Sections Immunohistochemically Stained to Detect Factor VIII (Von Willebrandt Factor)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: blood vessels/field
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 19 | 19
blood vessels/field | 4.9 (1.9) | 5.4 (2.2)

64. Secondary Outcome: Angiogenesis as Indicated by Number of Blood Vessels as Assessed by Light Microscopy of Biopsy Sections Immunohistochemically Stained to Detect Factor VIII (Von Willebrandt Factor)
Description: Gingival specimen biopsies (4mm in diameter, 1.5mm in thickness) will be harvested. The histological sections will be evaluated using a Nikon light microscope, and the area of angiogenesis will be quantified using Nikon NIS Element AR Imagine Software.
Time Frame: 10 days
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: blood vessels/field
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
Number analyzed (Participants) | 18 | 17
blood vessels/field | 4.4 (2) | 5.1 (2)

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Allogenic Amnion Chorion Membrane | Collagen Dressing
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03713073/Prot_SAP_000.pdf